CLINICAL TRIAL: NCT04448509
Title: Peripheral Blood Mononuclear Cell Collection Protocol for UCART Cell Tumor Immunotherapy Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: He Huang (Other)
Collaborators: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, He Huang, Clinical Professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BHCT-TCELL-04
Record Dates: First submitted 2020-06-19; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Peripheral Blood Mononuclear Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy donor (Other): Healthy donor
  Interventions: Other: Peripheral blood mononuclear cell apheresis

INTERVENTIONS:
Other: Peripheral blood mononuclear cell apheresis — Peripheral blood mononuclear cell collection for tumor immunotherapy study of UCAR-T cells

SUMMARY:
Peripheral blood mononuclear cell collection protocol for tumor immunotherapy study of UCAR-T cells

DETAILED DESCRIPTION:
Collect blood samples (whole blood and PBMC) from healthy donors for the development and production of UCAR-T cells

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-40 years, no donation reaction in the past;
2. Weight: male ≥ 50 kg, female ≥ 45 kg, and 18.5 kg/m2 ≤ BMI ≤ 30 kg/m2;
3. Blood pressure:12.0 Kpa (90 mmHg) ≤ systolic pressure﹤18.7 Kpa (140 mmHg) 8.0 Kpa (60 mmHg) ≤ diastolic pressure﹤12.0 Kpa (90 mmHg) Pulse pressure ≥ 4.0Kpa (30mmHg);
4. Pulse: 60/min to 100/min. Athletes with high endurance ≥ 50/min, with regular rhythm;
5. Temperature: 36.3-37.2℃ (oral temperature);
6. Generally in good condition: no damage to important organs such as heart, lung, liver and kidney; no severe or uncontrolled infection; no history of severe mental disorders;

Exclusion Criteria:

1. Valetudinarian, with frequent dizziness, giddiness, tinnitus, hemophobia, fear of needles, faint, and Meniere's disease;
2. Sexually transmitted diseases (STDs), leprosy, AIDS, and HIV-1, HIV-2, CMV, EBV antibody positive;
3. History of liver diseases, HBsAg positive and HCV antibody positive. 1 year after the clinical cure of hepatitis A, normal ALT test results at 1 month interval for 3 consecutive times;
4. Relapsed allergic diseases, urticaria, bronchial asthma and drug allergies (Donors with simple urticaria who are not in acute attack are eligible to donate PBMC);
5. Pulmonary tuberculosis, renal tuberculosis, lymph node tuberculosis and bone tuberculosis;
6. Urinary system diseases (e.g. acute and chronic nephritis, chronic urinary system infection, nephrotic syndrome, acute and chronic renal insufficiency, etc.);
7. Various hematological diseases (including anemia, leukemia, polycythemia vera and various hemorrhagic and coagulative diseases);
8. Endocrine diseases or metabolic disorders (e.g. hyperthyroidism, acromegaly, diabetes insipidus, diabetes mellitus, etc.);
9. Organic nervous system diseases or psychoses (e.g. encephalitis, sequelae of brain trauma, epilepsy, schizophrenia, hysteria, severe neurasthenia, etc.);
10. Parasitic diseases and endemic diseases (e.g. kala-azar, schistosomiasis, filariasis, hookworm disease, taeniasis, paragonimiasis, Keshan disease, Kaschin-Beck disease, etc.);
11. Malignancies and benign tumors affecting health;
12. Undergone resection of stomach, kidney, gallbladder, spleen, lung and other important organs;
13. Exposure to harmful substances or radioactive substances (except for clinical radiology);
14. High-risk groups susceptible to HIV infection, such as drug users, homosexuals and people with multiple sexual partners;
15. Creutzfeldt-Jakob disease (CJD), variant Creutzfeldt disease (vCJD), family history, and treatment with human and animal pituitary-derived substances (e.g. growth hormone, gonadotropin, thyrotropin, etc.). Organ transplantation recipients (including cornea, bone marrow, dura mater) may be exposed to bovine spongiform encephalopathy (BSE) and vCJD;
16. Other diseases or conditions in which donors are ineligible to donate PBMC in the opinion of physicians;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-07-18 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
the number of PBMC count | 1 years
  UCAR-T cell

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Zhejiang Medical Colleage Zhejiang University, Hangzhou, Zhejiang, China